CLINICAL TRIAL: NCT04341883
Title: A Open-label, Single-arm, Multicentre, Phase Ⅱ Study of Evaluate Efficacy and Safety of Anti-PD-1 Combined With Albumin-Bound Paclitaxel in Patients With Recurrent Cervical Cancer
Brief Title: Study of Anti-PD-1 Combined With Albumin-Bound Paclitaxel in Patients With Recurrent Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Hospital Chief Physician，Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-204-01
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Recurrent Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-PD-1 (Experimental): PD-1+albumin-bound paclitaxel
  Interventions: Drug: anti-PD-1+Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: anti-PD-1+Albumin-Bound Paclitaxel — anti-PD-1: 200mg/3w+Albumin-bound paclitaxel: 260 mg/m2/3w.Albumin-bound paclitaxel may be used for up to 6 cycles, and anti-PD-1 for up to 2 years.
  Other Name: Programmed cell death 1 antibody

SUMMARY:
This is an open-label, single-arm, phase II, multi-center clinical trial. Subjects can only enter this study after they meet the inclusion and exclusion criteria. All enrolled patients will receive the treatment with anti-PD-1 combined with albumin-bound paclitaxel, every 3 weeks, until progressive disease, initiation of new anti-tumour therapy, death, intolerable toxicity. Albumin-bound paclitaxel may be used for up to 6 cycles and anti-PD-1 for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and have signed the informed consent form (ICF);
2. Patients histologically diagnosed with cervical cancer ;
3. Patients with advanced cervical cancer who have experienced progressive disease or relapse after receiving standard treatment (first-line chemotherapy must be included) or who are intolerant to first-line chemotherapy.
4. The radiological examination during screening confirms the presence of at least one measurable lesion evaluated according to the RECIST v1.1;
5. An Eastern Cooperative Oncology Group(ECOG) score of 0 or 1;
6. Life expectancy ≥ 3 months;
7. Adequate hepatic, renal, heart, and hematologic functions. Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 70×109/L, Hemoglobin(HGB) ≥ 80 g/L, total bilirubin within 1.5×the upper limit of normal (ULN), and serum transaminase≤2.5×Upper Limit Of Normal(ULN), serum creatine ≤ 1.5 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥50ml/min, International Normalized Ratio<1.5 x Upper Limit Of Normal(ULN), Urinary protein≤（+）and Thyroid stimulating hormone≤ 1.5 x Upper Limit Of Normal(ULN).

Exclusion Criteria:

1. Pathology confirmed with sarcoma components (including malignant mixed mullerian tumors, endometrial leiomyosarcoma, and endometrial stromal sarcoma);
2. Patients who have previously received albumin-bound paclitaxel or exposures to any anti-PD-1 antibody drugs;
3. Exposures to any anti-tumor drugs within 4 weeks;
4. Current or prior use of any immunosuppressive medication or systemic hormone therapy（which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid Prednisone>10mg/d）within 14 days before the first dose of anti-PD-1 antibody;
5. Any primary malignancy within 5 years (except for fully treated in situ malignant such as breast cancer, bladder cancer, cervical carcinoma in situ, cutaneous basal cell carcinoma or squamous cell carcinoma);
6. History of psychiatric drugs abuse and not be abstinent, or dysphrenia；
7. Central nervous system diseases, including uncontrollable epilepsy and symptomatic brain metastases;
8. Severe cardiovascular disease: unstable angina pectoris, myocardial infarction, grade III-IV cardiac insufficiency (NYHA standard), and peripheral vascular disease above 2 degrees within 6 months prior to enrollment;
9. Severe arrhythmia requiring drug control, QT interval >470ms；
10. Active infections such as HIV/AIDS or other serious infectious diseases;
11. Any active autoimmune disease or history of autoimmune disease (including but not limit to autoimmune hepatitis, interstitial pneumonia, hepatitis, enteritis, nephritis, hyperthyroidism, pituitary inflammation, vasculitis, uveitis) . Patients need receiving systemic hormonal therapy and/or immunosuppressive therapy (eg asthma requiring bronchodilators);
12. Receipt of live attenuated vaccination within 30 days prior to study entry;
13. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 27 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 2 years
  Objective tumor response was defined as the proportion of patients whose tumor volume has been reduced to a predetermined value and can be maintained for more than 4 weeks, ie ORR=CR+PR.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | up to 2 years
  Progression-free survival was defined as the duration of time from study entry to time of progression, death, or the date of last contact, whichever occurs first.
Overall Survival(OS) | up to 2 years
  Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Disease Control Rate(DCR) | up to 2 years
  Disease control rate was defined as the proportion of subjects with complete response (CR) or partial response (PR) or disease stabilization (SD) in the analyzed population according to the RECIST 1.1 criteria.
Duration of Response(DoR) | up to 2 years
  Duration of response was defined as the time when the tumor is first evaluated as CR or PR to the first assessment for progressive disease(PD) or for any cause of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang Y, Zhao J, Liang H, Liu J, Huang S, Zou G, Huang X, Lan C. Efficacy and safety of sintilimab plus albumin-bound-paclitaxel in recurrent or metastatic cervical cancer: a multicenter, open-label, single-arm, phase II trial. EClinicalMedicine. 2023 Oct 24;65:102274. doi: 10.1016/j.eclinm.2023.102274. eCollection 2023 Nov. PMID 38106561